CLINICAL TRIAL: NCT02687763
Title: A Prospective, Multisite Study to Evaluate the Impact of Measles, Mumps, Rubella and Varicella ProQuad® Vaccination in Pediatric Patients 6-24 Months of Age Who Are Being Considered and/or Evaluated for Any Solid Organ Transplant
Brief Title: Safety and Efficacy of ProQuad® in Children 6-24 Month Being Evaluated for Solid Organ Transplant
Acronym: ProQuad®
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Katherine Twombley, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro25854
Record Dates: First submitted 2016-01-28; First posted 2016-02-22 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: RENAL INSUFFICIENCY, CHRONIC; LIVER FAILURE, ACUTE; HEART DISEASE
Keywords: vaccines; ProQuad; immunosuppressed; solid organ transplant; MMRV
MeSH Terms: conditions — Renal Insufficiency, Chronic; Liver Failure, Acute; Heart Diseases | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Open Label. Two 0.5-mL doses of ProQuad® will be given by intramuscular injection at least 30 days but no more than 365 days apart..
  Interventions: Biological: ProQuad

INTERVENTIONS:
Biological: ProQuad — 2) Patients 6 months to 24 months of age who are being considered and/or evaluated for any solid organ transplant within the next five (5) years who are willing:
  1. to receive two doses of ProQuad® at least 30 days but no more than 365 days apart.
  2. to participate in the three (3) antibody titer blood draws.

SUMMARY:
A prospective, multisite study to evaluate the Impact of Measles, Mumps, Rubella and Varicella ProQuad® vaccination in pediatric patients 6-24 months of age who are being considered and/or evaluated for any solid organ transplant (heart, liver or kidney)

DETAILED DESCRIPTION:
Primary Aim:

To measure the antibody response to ProQuad® vaccination given earlier than the current recommended age in patients from the age of 6 months to 24 months who are being considered and/or evaluated for any solid organ transplant (heart, liver or kidney) within the next five years. These subjects would not reach the recommended ages to receive the vaccine before the transplant.

Hypothesis:

The Investigator proposes the hypothesis that the proposed study population will mount a clinically significant response to two (2) doses of the ProQuad® vaccine.

Primary Endpoint:

With respect to expected outcomes, the work proposed is expected to provide tools for optimizing the ProQuad® vaccination strategy in this population.

Secondary Aim:

To determine the safety of ProQuad® vaccination in children aged 6 months to 24 months who are being considered and/or evaluated for any solid organ transplant (heart, liver, kidney).

Hypothesis :

The Investigator proposes the hypothesis that the study population will have similar safety profiles compared to children who receive the vaccine at the recommended ages.

Secondary Endpoint:

The secondary outcome measure is represented by the children in the study having either no adverse effects or minimal adverse effects from the ProQuad® vaccine. Adverse effects will be monitored via Electronic Medical Records (EMR) for Emergency Department (ED), hospital or clinic visits, follow-up phone calls to the family/subjects, as well as the vaccination report card that the parents/legal guardians of the participants in the study will complete for their child for 7 days after he/she receives each dose of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Parent and/or legal guardian willing and able to give informed consent.
2. Patients 6 months to 24 months of age who are being considered and/or evaluated for any solid organ transplant within the next five (5) years who are willing:

   * to receive two doses of ProQuad® at least 30 days but no more than 365 days apart.
   * to participate in the three (3) antibody titer blood draws.

Exclusion Criteria:

1. History of allergy to any vaccine component, bleeding disorder, exposure to measles, mumps, rubella, varicella, or zoster in the 30 days prior to vaccination.
2. Receipt of any blood product or immunoglobulin received in the previous 180 days prior to vaccination.
3. Previously received any measles, mumps, rubella and/or varicella vaccine either alone or in combination prior to vaccination.
4. Any condition which causes the investigator to determine that the subject is not appropriate to enroll.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

PRIMARY OUTCOMES:
Varicella IgG Antibody Titer ≥ 1.1 IU/ml | "at least 30 days to less than 365 days post vaccination"
  Percentage of Participants with Varicella IgG Antibody Titer ≥ 1.1 IU/ml: at least 30 days to less than 365 days post vaccination.
Measles IgG Antibody Titer ≥ 30AU/ml | "at least 30 days to less than 365 days post vaccination"
  Percentage of Participants with post vaccination Measles IgG Antibody Titer ≥ 30AU/ml: at least 30 days to less than 365 days post vaccination.
Mumps IgG Antibody Titer ≥ 11AU/ml | "at least 30 days to less than 365 days post vaccination"
  Percentage of Participants tested for Mumps IgG Antibody Titer ≥ 11AU/ml: at least 30 days to less than 365 days post vaccination.
Rubella IgG Antibody Titer ≥ 15 IU/mL | "at least 30 days to less than 365 days post vaccination"
  Percentage of Participants tested for Rubella IgG Antibody Titer ≥ 15 IU/mL: at least 30 days to less than 365 days post vaccination.

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Varicella Antibody | "at least 30 days to less than 365 days post vaccination"
  Geometric Mean Titer (GMT) of Varicella Antibody participating subjects at three different points in time. Antibody titers will be reported as geometric mean concentrations (GMCs) with 95% confidence intervals (CIs). Responses to historical controls will be compared by Student paired or unpaired t test and Fisher exact test. P < .05 will be considered statistically significant.
Geometric Mean Titer (GMT) of Measles Antibody | "at least 30 days to less than 365 days post vaccination"
  Geometric Mean Titer (GMT) of Measles Antibody participating subjects at three different points in time. Antibody titers will be reported as geometric mean concentrations (GMCs) with 95% confidence intervals (CIs). Responses to historical controls will be compared by Student paired or unpaired t test and Fisher exact test. P < .05 will be considered statistically significant.
Geometric Mean Titer (GMT) of Mumps Antibody | "at least 30 days to less than 365 days post vaccination"
  Geometric Mean Titer (GMT) of Mumps Antibody participating subjects at three different points in time. Antibody titers will be reported as geometric mean concentrations (GMCs) with 95% confidence intervals (CIs). Responses to historical controls will be compared by Student paired or unpaired t test and Fisher exact test. P < .05 will be considered statistically significant.
Geometric Mean Titer (GMT) of Rubella Antibody | "at least 30 days to less than 365 days post vaccination"
  Geometric Mean Titer (GMT) of Rubella Antibody participating subjects at three different points in time. Antibody titers will be reported as geometric mean concentrations (GMCs) with 95% confidence intervals (CIs). Responses to historical controls will be compared by Student paired or unpaired t test and Fisher exact test. P < .05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Twombley, MD, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Pediatric Nephrology, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No